CLINICAL TRIAL: NCT00751712
Title: Cerebral Oximetric Monitoring of the Posterior Circulation in Neonates and Infants During Complex Aortic Arch Reconstruction.
Brief Title: Cerebral Oximetric Monitoring of the Posterior Circulation
Acronym: CerebralOx
Status: Completed | Type: Observational
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 0511086
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Congenital Heart Disease
Keywords: Aortic Arch
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Back of skull cerebral oximeter sensor: All patients enrolled will receive non-invasive oxygen perfusion monitoring on the back of the skull during their standard of care congenital heart surgery
  Interventions: Device: Cerebral oximeter sensor

INTERVENTIONS:
Device: Cerebral oximeter sensor — The INVOS Cerebral Oximeter utilizes two electrodes to monitor cerebral oxygenation. The recommended placement of these electrodes is on the forehead to monitor the frontal cortex. In this study, one electrode will be placed in the normal position on the forehead, and the other will be placed at the base of the skull. The stickers will be placed on the patient at the beginning of surgery and removed at the end. The maximum amount of time that they will be on the patient's skin is approximately six hours. Application of the stickers and the data they provide will not alter the provider's treatment plan. This procedure will be used for all enrolled patients, whether they are enrolled in Part I or Part II.

SUMMARY:
One known risk of pediatric heart surgery is the possibility for brain damage. This problem results from a lack of oxygen rich blood flow to the brain during surgery. In order to provide the patient's brain with blood during this operation, selective cerebral perfusion is sometimes used. This technique allows for adequate blood flow to the brain, and is monitored using special sticker sensors. The sensors are applied to the patient's forehead, and a corresponding monitor indicates oxygen levels in the front part of the brain. The goal of this study is to find out if these same stickers can be applied to the base of the skull to measure cerebral oxygenation at the back of the brain, and to determine if the back of the brain is adequately oxygenated during selective cerebral perfusion in patients undergoing complex aortic arch reconstruction.

DETAILED DESCRIPTION:
One known risk of pediatric heart surgery is the possibility for brain damage. In may cases this problem results from a lack of oxygen rick blood flow to the brain during surgery. Recently, a technique has been developed that allows for adequate blood flow to the brain during surgery, thus decreasing the chances that brain injury will occur as a result of heart surgery. This technique, called selective cerebral perfusion, is not the technique of choice for surgeons operating to repair the aortic arch, but it is sometimes used. The aorta is the main artery that comes out of the heart and carries oxygen rick blood to the body. This large vessel is connected to the heart on one end and then extends upward and forms an arch. At the top of the arch, three vessels branch off and provide the upper part of the body, including the brain, with blood.

In a patient with a deformity in the aortic arch, it is necessary to operate to ensure that the flow of blood to the body is adequate and uninterrupted. In order to provide the baby's brain with blood during this operation, the technique mentioned earlier called selective cerebral perfusion is used. In order to understand how selective cerebral perfusion works, it is important to know that the patient will be placed on cardiopulmonary bypass during surgery. During cardiopulmonary bypass, a machine is used to pump blood to the body. This allows the surgeon to work on the heart and surrounding arteries while still providing blood flow of he brain and body. In the past, when surgery involved correction of abnormalities of the aortic arch, cardiopulmonary bypass would have to be stopped and the arch drained of blood, meaning there would be periods of time where the baby's brain would not receive any blood flow. With selective cerebral perfusion, a small Gore-Tex shunt is attached to one of the blood vessels that branch off of the aortic arch. Blood from the cardiopulmonary bypass machine is them pumped into the shunt where it enters the artery that branches off of the aorta and eventually travels up the neck and into the brain. Other studies have shown that pumping blood into this vessel allows the front portion of the brain to receive blood while the aortic arch abnormality is being corrected. These studies have shown this by using two stickers with special sensors on them that are connected to a monitor. These stickers, when placed on the baby's forehead, show on the monitor whether or not the front part of the brain is receiving blood.

There are two parts to this study, with part 1 used to assess feasibility:

Part 1: The goal of part one is to find out if these stickers can accurately show whether or not blood is getting to the back of the brain. Patients undergoing heart surgery who are not getting complex aortic arch reconstruction will be enrolled for part 1.

Part 2: If it is found that the stickers do work, part 2 will enroll patients who are undergoing complex aortic arch reconstruction. The goal of part 2 is to find out if the technique known as selective cerebral perfusion is effective at getting blood to the back of the brain during complex aortic arch reconstruction.

The study procedures for part 1 and 2 will be the same, with one sticker being placed in the normal position of the forehead, and the other sticker placed at the base of the skull. Application and data collected from the stickers in parts 1 and 2 will not affect surgical treatments.

ELIGIBILITY:
Inclusion Criteria:

Part I: Neonates or infants undergoing congenital heart surgery other than complex aortic arch reconstruction where surgical time is expected to be >= 1 hour in duration.

Part 2: Neonates or infants with complex aortic arch reconstruction where surgical time is expected to be >=1 hour in duration.

Exclusion Criteria:

* Neonates or infants with hydrocephalus
* Perinatal brain injury
* CNS (Central Nervous System) pathology, hemangiomas
* Cranial abnormalities
* Aortic or brachial anatomy that disallows performance of a shunt
* Skin conditions such as eczema or cradle cap.

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates or infants undergoing heart surgery
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2006-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Observational | Duration of Surgery

CONTACTS AND LOCATIONS:
Overall Officials: David M Overman, MD, Study Chair — Children's Heart Clinic
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No